CLINICAL TRIAL: NCT02077699
Title: Valutazione Dell'Efficacia Di Una Preparazione Commerciale A Base Di Lactobacillus Casei Dg Nella Riduzione Della Sintomatologia Dolorosa Associata Alla Sindrome Dell' Intestino Irritabile (Sii). Studio Clinico Pilota. (Official Title in Italian Language)
Brief Title: Efficacy Evaluation of a Commercial Preparation Containing Lactobacillus Casei DG on the Reduction of the Painful Symptoms Related to the Irritable Bowel Syndrome (IBS). A Pilot Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBS-DG 10
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Lactobacillus casei DG; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment with Lactobacillus casei DG (24 billion of live cells per pill) 2 pills b.i.d. for 4 weeks
  Interventions: Dietary Supplement: Lactobacillus casei DG

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei DG — Lactobacillus casei DG (24 billion of live cells per pill) - 2 pills b.i.d. for 4 weeks
  Other Names: Enterolactis plus

SUMMARY:
The purpose of this study is to evaluate the efficacy of a treatment with Lactobacillus casei DG in the reduction of the painful symptoms in patients affected by irritable bowel syndrome. After that, the secondary object is to evaluate if the reduction of painful symptoms is related to a relevant reduction of trypsin and tryptase in colonic mucosa.

ELIGIBILITY:
Inclusion Criteria:

* out-Patients with diagnosis of Irritable Bowel syndrome (IBS) according to Rome III Diagnostic Criteria for Functional Gastrointestinal Disorders
* Previous colonoscopy (within 24 month prior the enrollment) with negative results
* written informed consent

Exclusion Criteria:

* systemic or topical therapy with steroids and glucocorticoids such as beclomethasone dipropionate or budesonide, ongoing or within a month prior the enrollment
* therapy with antibiotics or probiotics, ongoing or within a month prior the enrollment
* inflammatory bowel diseases
* copro-paraxitological examination with positive results
* bowel disease with infectious, actinic, endocrine or drug-related origin
* immunodeficiency
* diagnosis of malignant cancer within 5 years prior the enrollment
* renal, hepatic, hematologic, cardiovascular, pulmonary, neurological, psychiatric, immunological, gastrointestinal or endocrine disorders, if found to be clinically relevant
* any severe disease that may interfere with the treatment;
* abuse of alcohol, drugs or medication, psychotropic drugs
* diagnosis of dementia or other disorders that can cause a progressive deterioration of capacity of discernment or mental and physical disability which reduces the ability to follow the prescribed therapy;
* previous participation in this study
* pregnant or nursing (lactating) women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Intensity of painful symptoms | 4 weeks
  The efficacy of the treatment will be evaluated recording the intensity of the painful symptoms associated with irritable bowel syndrome for the duration of the study. The intensity of abdominal pain will be recorded daily by the patient in a diary using a semi-quantitative scale (Likert) to 6 points, from 0 (absent) to 5 (very severe).

SECONDARY OUTCOMES:
Level of trypsin and tryptase in colonic mucosa | 4 weeks
  Will evaluate the reduction in the levels of trypsin and tryptase in the colonic mucosa by collecting biopsies from the sigmoid colon and samples colonic lavage fluid and subsequent histological and molecular examination with extraction of m-RNA and proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Monteleone, Professor, Principal Investigator — Policlinico Tor Vergata
Locations (1):
- UOC di Gastroenterologia - Policlinico Tor Vergata, Roma, Roma, Italy

REFERENCES:
- [Background] Hungin AP, Chang L, Locke GR, Dennis EH, Barghout V. Irritable bowel syndrome in the United States: prevalence, symptom patterns and impact. Aliment Pharmacol Ther. 2005 Jun 1;21(11):1365-75. doi: 10.1111/j.1365-2036.2005.02463.x. PMID 15932367
- [Background] Thompson WG, Longstreth GF, Drossman DA, Heaton KW, Irvine EJ, Muller-Lissner SA. Functional bowel disorders and functional abdominal pain. Gut. 1999 Sep;45 Suppl 2(Suppl 2):II43-7. doi: 10.1136/gut.45.2008.ii43. PMID 10457044
- [Background] Langhorst J, Junge A, Rueffer A, Wehkamp J, Foell D, Michalsen A, Musial F, Dobos GJ. Elevated human beta-defensin-2 levels indicate an activation of the innate immune system in patients with irritable bowel syndrome. Am J Gastroenterol. 2009 Feb;104(2):404-10. doi: 10.1038/ajg.2008.86. Epub 2009 Jan 20. PMID 19174795
- [Background] Salzmann JL, Peltier-Koch F, Bloch F, Petite JP, Camilleri JP. Morphometric study of colonic biopsies: a new method of estimating inflammatory diseases. Lab Invest. 1989 Jun;60(6):847-51. PMID 2733385
- [Background] O'Sullivan M, Clayton N, Breslin NP, Harman I, Bountra C, McLaren A, O'Morain CA. Increased mast cells in the irritable bowel syndrome. Neurogastroenterol Motil. 2000 Oct;12(5):449-57. doi: 10.1046/j.1365-2982.2000.00221.x. PMID 11012945
- [Background] Barbara G, Stanghellini V, De Giorgio R, Cremon C, Cottrell GS, Santini D, Pasquinelli G, Morselli-Labate AM, Grady EF, Bunnett NW, Collins SM, Corinaldesi R. Activated mast cells in proximity to colonic nerves correlate with abdominal pain in irritable bowel syndrome. Gastroenterology. 2004 Mar;126(3):693-702. doi: 10.1053/j.gastro.2003.11.055. PMID 14988823
- [Background] Gwee KA, Collins SM, Read NW, Rajnakova A, Deng Y, Graham JC, McKendrick MW, Moochhala SM. Increased rectal mucosal expression of interleukin 1beta in recently acquired post-infectious irritable bowel syndrome. Gut. 2003 Apr;52(4):523-6. doi: 10.1136/gut.52.4.523. PMID 12631663
- [Background] Fahlgren A, Hammarstrom S, Danielsson A, Hammarstrom ML. beta-Defensin-3 and -4 in intestinal epithelial cells display increased mRNA expression in ulcerative colitis. Clin Exp Immunol. 2004 Aug;137(2):379-85. doi: 10.1111/j.1365-2249.2004.02543.x. PMID 15270856
- [Background] O'Mahony L, McCarthy J, Kelly P, Hurley G, Luo F, Chen K, O'Sullivan GC, Kiely B, Collins JK, Shanahan F, Quigley EM. Lactobacillus and bifidobacterium in irritable bowel syndrome: symptom responses and relationship to cytokine profiles. Gastroenterology. 2005 Mar;128(3):541-51. doi: 10.1053/j.gastro.2004.11.050. PMID 15765388
- [Background] Rembacken BJ, Snelling AM, Hawkey PM, Chalmers DM, Axon AT. Non-pathogenic Escherichia coli versus mesalazine for the treatment of ulcerative colitis: a randomised trial. Lancet. 1999 Aug 21;354(9179):635-9. doi: 10.1016/s0140-6736(98)06343-0. PMID 10466665
- [Background] Venturi A, Gionchetti P, Rizzello F, Johansson R, Zucconi E, Brigidi P, Matteuzzi D, Campieri M. Impact on the composition of the faecal flora by a new probiotic preparation: preliminary data on maintenance treatment of patients with ulcerative colitis. Aliment Pharmacol Ther. 1999 Aug;13(8):1103-8. doi: 10.1046/j.1365-2036.1999.00560.x. PMID 10468688